CLINICAL TRIAL: NCT03482167
Title: NAD Therapy for Improving Memory and Brain Blood Flow in Older Adults With Mild Cognitive Impairment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christopher Martens, Assistant Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1079271; K01AG054731 (NIH)
Record Dates: First submitted 2018-02-14; First posted 2018-03-29 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment
Keywords: blood pressure; arterial stiffness; cerebrovascular function; cognitive function
MeSH Terms: conditions — Cognitive Dysfunction | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Other: Placebo
- Nicotinamide Riboside (Experimental): Niagen® (ChromaDex, Inc.) 500 mg, twice daily
  Interventions: Drug: Niagen®

INTERVENTIONS:
Drug: Niagen® — 250 mg capsules (4 capsules daily)
  Other Names: nicotinamide riboside chloride
  Arms: Nicotinamide Riboside
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
This study will provide insight into whether a nutritional supplement, nicotinamide riboside (NR), improves memory and brain blood flow in older adults with low memory abilities. Overall, this project has the potential to identify a novel, safe and cost-effective strategy for decreasing age-related memory loss.

ELIGIBILITY:
Inclusion Criteria

* Cognitive function scores consistent with amnestic mild cognitive impairment based on pre-screening evaluation;
* age 60-90 years;
* MMSE score >24 at time of initial consent;

Exclusion Criteria

* blood chemistries indicative of abnormal renal, liver, thyroid and adrenal function; estimated glomerular filtration rate using the MDRD prediction equation must be >30 ml/min/1.73 m2;
* any clinically significant abnormal blood chemistry values as determined by the research nurse or NMPCC nurse practitioner;
* major psychiatric disorder (e.g. schizophrenia, bipolar disorder, major depression within past two years);
* neurological or autoimmune conditions affecting cognition (e.g. Parkinson's disease, epilepsy, multiple sclerosis, mild or severe traumatic brain injury, large vessel infarct);
* concussion within last 2 years and ≥ 3 lifetime concussions;
* current systemic medical illnesses (e.g. cardiovascular disease, cancer, renal failure);
* prior history of any type of cancer;
* substance abuse or dependence (DSM-V criteria);
* current use of medications used to treat dementia (e.g., anticholinesterase drugs) or other drugs likely to affect cognition (e.g., anticholinergic drugs, long-acting benzodiazepines);
* claustrophobia, metal implants, pacemaker or other factors affecting feasibility and/or safety of MRI scanning*;
* current smoking (including marijuana) within the past 3 months;
* hospitalization as a result of COVID-19

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Martens, Ph.D., Principal Investigator — University of Delaware
Locations (1):
- Neurovascular Aging Laboratory, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened for inclusion in this study at the University of Delaware between March 20, 2019 - August 21, 2023.
Pre-assignment Details: A total of 64 participants were consented into this study. Of these, 13 participants were withdrawn prior to randomization. Reasons for withdrawal inlcluded not meeting eligibility criteria (N = 7), failure to comply with study requirements (N = 1), voluntarily withdrawal by the participant (N = 2), or if a participant was lost to followup (N = 2).
Period: Allocated to Intervention
Arm/Group | Placebo | Nicotinamide Riboside
Started | 26 | 26
Completed | 25 | 24
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 2
Period: Received Intervention
Arm/Group | Placebo | Nicotinamide Riboside
Started | 25 | 24
Completed | 20 | 22
Not Completed | 5 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Criteria for amnestic mild cognitive impairment (MCI) included lack of dementia and at least one memory score ≤ 1.5 standard deviations from the mean.
  One (1) participant allocated to placebo was withdrawn prior to treatment due to disclosure of prior cancer history, which was a stated exclusion criterion.
  Two (2) participants allocated to NR were withdrawn prior to starting treatment due to disclosure of prior cancer history, which was a stated exclusion criterion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nicotinamide Riboside | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (7) | 72 (8) | 72 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 24 | 23 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 16 | 22 | 38
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
APOE ε4 Carrier [Count of Participants; unit: Participants] — One or more copy of the APOE ε4 allele
  Participants | 10 | 10 | 20
APOE Genotype [Count of Participants; unit: Participants]
  ε2/ε2 | 0 | 0 | 0
  ε2/ε3 | 6 | 4 | 10
  ε2/ε4 | 2 | 0 | 2
  ε3/ε3 | 9 | 10 | 19
  ε3/ε4 | 8 | 9 | 17
  ε4/ε4 | 0 | 1 | 1
Mini Mental State Exam (MMSE) [Mean (Standard Deviation); unit: Units on a scale] — Total Score on the MMSE ranges between 0-30, with a higher score indicative of better cognitive function. A Total Score below 20 is indicative of moderate to severe dementia and was used a cutoff for inclusion in this study.
  Units on a scale | 27 (2) | 26 (2) | 27 (2)
Clinical Dementia Rating - Global Score [Mean (Standard Deviation); unit: units on a scale] — The Global Clinical Dementia Rating (CDR) Score is a calculated weighted score derived from the following six "box scores": 1) Memory, 2) Orientation, 3) Judgment and problem-solving, 4) Community affairs, 5) Home and hobbies, and 6) Personal care. Global CDR Score is used to assess level of impairment and severity of dementia based on the following scale:
  0 = Normal; 0.5 = Very Mild Dementia; 1 = Mild Dementia; 2 = Moderate Dementia; 3 = Severe Dementia
  units on a scale | 0.4 (0.2) | 0.4 (0.2) | 0.4 (0.2)
Revised Hopkins Verbal Learning Test (HVLT-R) Total Recall Memory [Mean (Standard Deviation); unit: T-Score] — The Revised Hopkins Verbal Learning Test (HVLT-R) assesses verbal learning and memory, immediate recall, delayed recall, and delayed recognition. Total Recall T-score was used in the determination of mild cognitive impairment (MCI). A T-score of 50 represents the population mean with a standard deviation of 10. A T-score <50 indicates below average cognitive function and a T-score ≤ 35 is potentially indicative of MCI.
  T-Score | 39 (8) | 38 (8) | 39 (8)
Revised Brief Visuospatial Memory Test (BVMT-R) Total Recall Score [Mean (Standard Deviation); unit: T-Score] — The Revised Brief Visuospatial Memory Test (BVMT-R) assesses visuospatial memory and includes an immediate and delayed recall. Total Recall T-score was used in the determination of mild cognitive impairment (MCI). A T-score of 50 represents the population mean with a standard deviation of 10. A T-score <50 indicates below average cognitive function and a T-score ≤ 35 is potentially indicative of MCI. Population: Screening for MCI status occurred in-person until March 2020 when the study was temporarily stopped due to the COVID-19 pandemic. Prior to the pandemic, we used the BVMT, in-person, in our screening pipeline for MCI status. After the pandemic, we began doing most of our screenings using online video conferencing. Because the BVMT cannot easily be administered online, we switched to using the WMS Logical Memory Test.
  T-Score
    number analyzed (Participants) | 4 | 8 | 12
    (all) | 35 (13) | 33 (8) | 35 (8)
Revised Wechsler Memory Scale (WMS-R) - Logical Memory I [Mean (Standard Deviation); unit: units on a scale] — The Logical Memory I (immediate recall) is a subset of the Wechsler Memory Scale and assesses the ability to immediately recall aspects of a story. Scaled scores range from 1-19 and are derived from 100 normative cases within a specific age band. The scaled score is based on a normal distribution with a mean of 10 and a standard deviation of 3. A scaled score of at least 1.5 standard deviations below the mean is potentially indicative of MCI. Population: Screening for MCI status occurred in-person until March 2020 when the study was temporarily stopped due to the COVID-19 pandemic. Prior to the pandemic, we used the BVMT, in-person, in our screening pipeline for MCI status. After the pandemic, we began doing most of our screenings using online video conferencing. Because the BVMT cannot easily be administered online, we switched to using the WMS Logical Memory Test.
  units on a scale
    number analyzed (Participants) | 21 | 16 | 37
    (all) | 8 (3) | 8 (3) | 8 (3)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Scores at Baseline and Week 12
Description: Primary outcome was a change from baseline in any domain of cognitive function. For all outcomes, a higher score indicates better cognitive function:
  1. California Verbal Learning Test III (CVLT-III) Index Scores. Ability learn and recall a list of words over 5 trials and again after a 20 minute delay. Each Index Score has a mean of 100 and a standard deviation of 15 based on normative dataset (Range = 55 - 145).
  2. Wechsler Memory Scale IV (WMS-IV) Raw Scores.
     * Logical Memory I & II: Range = 0-50
     * Logical Memory II Recognition: Range = 0-30
     * Visual Reproduction I & II: Range = 0-43
     * Visual Reproduction II Recognition Score: Range = 0-7
  3. NIH Toolbox Fluid Composite Score. Composite Score has a mean of 100 and a standard deviation of 15 based on normative dataset (Range = 55 - 145) - based on several tests of fluid and crystallized cognition (episodic memory, attention, working memory, processing speed, executive function and language abilities).
Time Frame: baseline and 12 weeks
Population: Number of cases analyzed for select cognitive tests differs from overall number analyzed due to missing data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Nicotinamide Riboside
Number analyzed (Participants) | 20 | 22
score on a scale
  CVLT3 Trial 1-5 Index Score (Baseline) | 96 (4) | 99 (4)
  CVLT3 Trial 1-5 Index Score (Week 12): number analyzed (Participants) | 20 | 21
  CVLT3 Trial 1-5 Index Score (Week 12) | 101 (3) | 103 (4)
  CVLT3 Delayed Recall Index Score (Baseline) | 93 (3) | 93 (4)
  CVLT3 Delayed Recall Index Score (Week 12): number analyzed (Participants) | 20 | 21
  CVLT3 Delayed Recall Index Score (Week 12) | 97 (4) | 100 (4)
  CVLT3 Total Recall Index Score (Baseline) | 95 (4) | 96 (4)
  CVLT3 Total Recall Index Score (Week 12): number analyzed (Participants) | 20 | 21
  CVLT3 Total Recall Index Score (Week 12) | 99 (3) | 101 (4)
  WMS-IV Logical Memory I Total Raw Score (Baseline) | 18 (1) | 20 (2)
  WMS-IV Logical Memory I Total Raw Score (Week 12): number analyzed (Participants) | 20 | 21
  WMS-IV Logical Memory I Total Raw Score (Week 12) | 21 (1) | 25 (2)
  WMS-IV Logical Memory II Total Raw Score (Baseline) | 15 (1) | 15 (2)
  WMS-IV Logical Memory II Total Raw Score (Week 12): number analyzed (Participants) | 20 | 21
  WMS-IV Logical Memory II Total Raw Score (Week 12) | 16 (2) | 19 (2)
  WMS-IV Logical Memory II Recognition Total Raw Score (Baseline) | 23 (1) | 22 (1)
  WMS-IV Logical Memory II Recognition Total Raw Score (Week 12): number analyzed (Participants) | 20 | 21
  WMS-IV Logical Memory II Recognition Total Raw Score (Week 12) | 23 (1) | 24 (1)
  WMS-IV Visual Reproduction I Total Raw Score (Baseline) | 29 (1) | 29 (2)
  WMS-IV Visual Reproduction I Total Raw Score (Week 12) | 30 (2) | 30 (2)
  WMS-IV Visual Reproduction II Total Raw Score (Baseline) | 17 (2) | 17 (2)
  WMS-IV Visual Reproduction II Total Raw Score (Week 12) | 19 (2) | 18 (2)
  WMS-IV Visual Reproduction II Recognition Total Raw Score (Baseline) | 5 (0.001) | 5 (0.001)
  WMS-IV Visual Reproduction II Recognition Total Raw Score (Week 12) | 6 (0.001) | 5 (0.001)
  NIH Toolbox Fluid Cognition Score (Baseline): number analyzed (Participants) | 20 | 21
  NIH Toolbox Fluid Cognition Score (Baseline) | 87 (2) | 84 (3)
  NIH Toolbox Fluid Cognition Score (Week 12) | 89 (3) | 84 (3)

2. Secondary Outcome: Cerebrovascular Reactivity at Baseline and 12 Weeks
Description: Relative (percent) change in blood velocity of the middle cerebral artery (MCA) per mmHg change in end-tidal carbon dioxide (ETCO2) during a brief period of hypercapnia.
  Hypercapnia was induced by prospective end-tidal targeting (RespirAct, Thornhill Medical) in which a target change in end-tidal CO2 of +9mmHg was set. Data were only analyzed if ETCO2 changed by at least 6mmHg. All data were then normalized to the absolute change in ETCO2.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: % change in MCAv (m/sec) per mmHg ETCO2
Arm/Group | Placebo | Nicotinamide Riboside
Number analyzed (Participants) | 2 | 5
% change in MCAv (m/sec) per mmHg ETCO2
  Percent change in MCA velocity per mmHg change in ETCO2 - Baseline | 3.2 (1.9) | 1.1 (1.0)
  Percent change in MCA velocity per mmHg change in ETCO2 - Week 12 | 4.2 (0.8) | 2.8 (0.7)

3. Secondary Outcome: Total Brain Blood Flow at Baseline and 12 Weeks
Description: Total brain blood flow assessed by pseudo-continuous arterial spin labeling (pcASL). Total brain blood flow is measured in milliliters of blood per minute per 100 grams of brain tissue.
Time Frame: baseline and 12 weeks
Population: Number of cases analyzed for select cognitive tests differs from overall number analyzed due to missing data.
Measure: Mean (Standard Error); unit: ml/min/100g
Arm/Group | Placebo | Nicotinamide Riboside
Number analyzed (Participants) | 20 | 22
ml/min/100g
  Baseline: number analyzed (Participants) | 17 | 19
  Baseline | 47.1 (2.9) | 48.6 (4.3)
  Week 12: number analyzed (Participants) | 17 | 18
  Week 12 | 47.4 (2.7) | 55.5 (4.0)

4. Secondary Outcome: Aortic Stiffness at Baseline and 12 Weeks
Description: Carotid-femoral pulse wave velocity (CFPWV)
Time Frame: baseline and 12 weeks
Population: Number of cases analyzed for select cognitive tests differs from overall number analyzed due to missing data.
Measure: Mean (Standard Error); unit: m/sec
Arm/Group | Placebo | Nicotinamide Riboside
Number analyzed (Participants) | 20 | 22
m/sec
  Baseline: number analyzed (Participants) | 19 | 21
  Baseline | 8.9 (0.4) | 9.8 (0.4)
  Week 12: number analyzed (Participants) | 18 | 21
  Week 12 | 8.5 (0.5) | 9.1 (0.5)

5. Secondary Outcome: Blood Pressure at Baseline and 12 Weeks
Description: Seated systolic and diastolic blood pressure assessed using automated oscillometric sphygmomanometer.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Nicotinamide Riboside
Number analyzed (Participants) | 20 | 22
mmHg
  Systolic (Baseline) | 124 (3) | 132 (3)
  Systolic (Week 12) | 123 (3) | 127 (3)
  Diastolic (Baseline) | 70 (2) | 74 (2)
  Diastolic (Week 12) | 72 (2) | 73 (2)

6. Other Pre Specified Outcome: Neurovascular Coupling at Baseline and 12 Weeks
Description: Cerebrovascular reactivity to cognitive tasks
Time Frame: baseline and 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Functional Brain Connectivity at Baseline and 12 Weeks
Description: functional brain connectivity assessed by MRI
Time Frame: baseline and 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Neuronal Activation at Baseline and 12 Weeks
Description: Functional MRI (fMRI) to cognitive task
Time Frame: baseline and 12 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Brain Volume at Baseline and 12 Weeks
Description: White and grey matter volume assessed by structural MRI
Time Frame: baseline and 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Nicotinamide Riboside
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 12/25 | 8/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Nicotinamide Riboside (N=24)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Poison Ivy
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0) — Sleep disturbance
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Heart palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — panic attack
Triglycerides increased (Investigations) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Technical problems with ultrasound measures leading to unreliable or uninterpretable data in some participants. Total brain blood flow was therefore assessed in all participants by MRI using pseudo-continuous arterial spin labeling (pCASL).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT03482167/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03482167/ICF_001.pdf